CLINICAL TRIAL: NCT05211752
Title: Eye Movements Recording Using a Smartphone: Comparison to Standard Video-oculography Data in Young Athletes
Brief Title: Eye Movements Recording Using a Mobile : Comparison to Standard Video-oculography in Young Athletes
Acronym: e-VOG(YA)
Status: Completed | Type: Observational
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other); Centre Hospitalier Universitaire de Nice (Other); Association Sportive Monaco Football Club (Unknown)
Responsible Party: Sponsor
Other Study IDs: e-VOG Young Athletes
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Young Athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy young athletes (Eye-Tracker®T2 + e-VOG): Subjects who first perform standard video-oculography assessment, followed by e-VOG digital assessment.
  Interventions: Other: eVOG (Mobile VideoOculoGraphy)
- Healthy young athletes (e-VOG + Eye-Tracker®T2): Subjects who first perform e-VOG digital assessment, followed by the standard video-oculography assessment.
  Interventions: Other: eVOG (Mobile VideoOculoGraphy)

INTERVENTIONS:
Other: eVOG (Mobile VideoOculoGraphy) — * Eyes movements assessed with e-VOG (mobile application, that uses the face detection features of the front camera to detect and record eye movements).
  * Study duration is about 20 minutes, the day the subject performs his standard video-oculography examination in routine care (using Eye-Tracker®T2)

SUMMARY:
This study aims to compare measurements obtained through the e-VOG application (mobile application, usable on smartphones or tablets, to measure eye movements) with measurements from the standard video-oculography device (Eye-Tracker®T2), in young athletes.

DETAILED DESCRIPTION:
e-VOG Young athletes is a collaborative study between the Memory Center of the Rainier III Center (Princess Grace Hospital, Monaco), the Neurology Department of Nice University Hospital (France), and the AS Monaco Football Academy medical team.

Memory Center of the Rainier III Center is expert in eye-tracking and is equipped with a standard video-oculography device (Eye-Tracker®T2), which records eye movements at a high frequency and measures saccades parameters (latency, speed, amplitudes etc...).

e-VOG is a mobile application, home-developed by the Neurology Department team of Nice University Hospital, to measure eye movements.

Based on literature, investigators hypothesize that video-oculography could integrate assessment protocols for head trauma occurring during sports practice. The nomadic nature of the e-VOG application would make possible to assess oculomotor behaviors to a subject who has just suffered a trauma and who is suspected of having a concussion.

From this perspective, it seems necessary to firstly validate baseline values of the e-VOG application in a population of athletes without major health problems, and who have not presented concussion.

ELIGIBILITY:
Inclusion Criteria:

* Young Athletes from AS Monaco Football Academy
* referred by AS Monaco Medical Team to perform a video-oculography (Eye-Tracking) examination as part of routine care.
* covered by a health insurance system
* volunteer, able to give free, informed and written consent.
* For minors: whose holder of parental authority has given their written consent to participate following the information given by investigator.

Exclusion Criteria:

* General anaesthesia within 3 months.
* Head trauma within 3 months
* Neurological, ophthalmological or general pathology preventing the realization of a video-oculography examination.
* Oculomotor abnormality detectable on clinical examination by the neurologist prescribing the standard video-oculography examination.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young athletes for whom a standard video-oculography exam is prescribed by the AS Monaco Football medical team as part of a preventive and follow-up approach performed in routine care.
  Eye-tracking is a relevant and essential assessment for the detection and monitoring of neuro-cognitive alterations in young athletes which may result from macro-trauma (concussion) or repeated micro-trauma (head game) occurring during the season.
  Standard video-oculography exam is carried out at the Center Rainier III (Princess Grace Hospital), in accordance with usual practices. It is a non-invasive device for eye movements recording, allowing doctors to measure standard parameters related to eye movements (Class IIa medical device, CE marking, according to Annexe IX of the directive 93/42/CE).
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Oculomotor profiles concordance | Day 0
  Analyze of the concordance of the profiles obtained between the e-VOG digital assessment and the standard video-oculography assessment.
  Evaluation criteria: For each assessment, patients will be classified according to the number of oculomotor abnormality observed (based on identified parameters assessments: latency / speed / gain / altered ocular pursuits / fixation disorders / presence of internuclear ophthalmoplegia), in accordance with the literature standards.

SECONDARY OUTCOMES:
Latency during horizontal reflex saccades | Day 0
  Measure of Latency during an horizontal reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Latency during vertical reflex saccades | Day 0
  Measure of Latency during a vertical reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Latency during horizontal voluntary saccades | Day 0
  Measure of Latency during an horizontal volontary saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Velocity during horizontal reflex saccades | Day 0
  Measure of Velocity during an horizontal reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: velocity (mean and peak velocity) in °/s.
Velocity during vertical reflex saccades | Day 0
  Measure of Velocity during a vertical reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: velocity (mean and peak velocity) in °/s.
Inhibition capacity | Day 0
  Measure of inhibition capacity performance during an antisaccades" paradigm with e-VOG Compared to the one evaluated with standard video-oculography device.
  Evaluation criteria: percentage of errors.
Internuclear ophthalmoplegia (INO) detection | Day 0
  Highlight presence/absence of INO with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: INO is present if calculated ratio of abducting to adducting eye movement (both mean and peak velocity) is >1.
Fixations impairments detection | Day 0
  Highlight presence/absence of Fixations impairments with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence/frequency of square wave-jerks, nystagmus, flutters.
Impairment of horizontal smooth pursuit | Day 0
  Highlight Impairment of horizontal smooth pursuit with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence of saccade and perturbation.
Impairment of vertical smooth pursuit | Day 0
  Highlight Impairment of horizontal smooth pursuit with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence of saccade and perturbation.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael COHEN, MD, Principal Investigator — Centre de Ressources et de Compétences SEP, UMRC Pasteur 2, Université Nice Côte d'Azur, Nice-France; Sandrine LOUCHART de la CHAPELLE, MD-PHD, Principal Investigator — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital, Monaco; Alain PESCE, PUPH, Study Director — Association de Recherche Bibliographique pour les Neurosciences; Sylvain BLANCHARD, MD-PHD, Principal Investigator — Association Sportive Monaco Football Club
Locations (1):
- Centre Mémoire / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No